CLINICAL TRIAL: NCT01201083
Title: Transmission Behavior in Partnerships of Newly HIV Infected Southern Californians
Brief Title: Study of Recently HIV Infected Men and Transmission Behaviors
Acronym: MetroMates
Status: Completed | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Collaborators: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Responsible Party: Principal Investigator, Pamina Gorbach, Principal Investigator, University of California, Los Angeles
Other Study IDs: R01DA022116 - A1; G07-06-117-03 (Other: UCLA); R01DA022116 (NIH)
Record Dates: First submitted 2010-09-09; First posted 2010-09-14 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: HIV

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — We collect a sample of blood/plasma and have a repository (blood) and for future analysis. After noting that subject has consented to main study as well as consenting to have his blood stored for later research purposes, appropriate research staff will direct the phlebotomist to draw and additional tube of blood (approximately 7mls of blood) into a purple cap (EDTA) tube. After processing, each sample will be securely stored at the participating site under appropriate conditions .
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- HIV-: This study measured how transmission risks and partnership dynamics change over time among recently HIV-infected individuals and their partners comparing their behavioral patterns with those with chronic HIV infection, no HIV infection, and HIV negative testers. Of special focus was the role of drug use, especially methamphetamine, in affecting behaviors over time, and how partnership dynamics interact with drug use to allow for HIV transmission. The study compared behaviors of recently HIV infected men to those with long-term HIV infection and no HIV infection. We looked at how different types of sex partners affected one's drug use and consequently HIV transmission risks including having a prevalent sexually transmitted infection (STI). The study enrolled 105 HIV- recently tested men who have sex with men (MSM) and followed them for a year.
- HIV+ Acutely Infected: This study enrolled and followed 125 acutely infected HIV+ men. It measured how transmission risks and partnership dynamics change over time among recently HIV-infected individuals and their partners comparing their behavioral patterns with those with chronic HIV infection, no HIV infection, and HIV negative testers. Of special focus was the role of drug use, especially methamphetamine, in affecting behaviors over time, and how partnership dynamics interact with drug use to allow for HIV transmission. The study compared behaviors of recently HIV infected men to those with long-term HIV infection and no HIV infection. We looked at how different types of sex partners affected one's drug use and consequently HIV transmission risks including having a prevalent sexually transmitted infection (STI). The study enrolled 321 recently tested men who have sex with men (MSM) and followed them for a year.
- HIV+ Chronically Infected: This study enrolled and followed 91chronicially infected HIV+ men. It measured how transmission risks and partnership dynamics change over time among recently HIV-infected individuals and their partners comparing their behavioral patterns with those with chronic HIV infection, no HIV infection, and HIV negative testers. Of special focus was the role of drug use, especially methamphetamine, in affecting behaviors over time, and how partnership dynamics interact with drug use to allow for HIV transmission. The study compared behaviors of recently HIV infected men to those with long-term HIV infection and no HIV infection. We looked at how different types of sex partners affected one's drug use and consequently HIV transmission risks including having a prevalent sexually transmitted infection (STI). The study enrolled 321 recently tested men who have sex with men (MSM) and followed them for a year.

SUMMARY:
Identify drug use patterns and partnership dynamics that mediate risk behaviors over time in a cohort of recently HIV infected men and their partners; to determine predictors of transmission risk within partnerships of recently HIV infected men and their partners, using the partnership as the unit of analysis; and to quantify the long-term population-level impacts of voluntary behavior change by men with recent HIV infection, through the use of dynamic mathematical modeling that integrates our data on behavior change with current estimates of temporal infectiousness patterns. The investigators will also determine whether more frequent testing and/or development of tests with earlier sensitivity may have a significant impact on the epidemic. Finally, the magnitude of this effect to that obtained by decreasing drug use or risky sexual behavior prior to or following seroconversion will be compared. This will be conducted as a statistical analysis by co-investigators at the University of Washington.

DETAILED DESCRIPTION:
People who recently became infected with HIV often have a high level of the virus and may be highly infectious. If they have sex (especially anal intercourse) without condoms soon after they have been infected with HIV, there is a great chance that they may transmit the virus to others. When they learn of their HIV infection, some but not all men change sexual behaviors so as not to infect their partner(s) with HIV. Possible reasons for such behavior change include increase or decrease in drug use and what is going on within their sexual partnerships. A study that tracks men with recent HIV infection and their partners over time can provide information key to stopping further spread of HIV given that sexual behaviors can vary over time, especially during this most infectious period.

This study will look at how likely it is for HIV infection to be spread among partner types over time by recently HIV-infected men and their partners. The study will compare behaviors of recently HIV infected men to those with long-term HIV infection and no HIV infection. It will allow a study of sexual partnerships by actively recruiting sexual partners. We will also focus on the role of drug use, especially methamphetamine and how it changes behaviors over time. We will especially look at how different sex partners affects one's drug use and increases or decreases HIV transmission. The study will enroll 150 recently HIV-infected men who have sex with men and follow them for a year. In addition, up to 6 sexual partners of each recently HIV infected individual will be recruited and followed for a year. Some sexual partners will be HIV negative and some HIV positive. We will use their HIV status to compare behaviors over time in the group and between partners of the same status and partners of a different status. The results will be used in special formulas that will allow for a better understanding of behavior change by men with recent HIV infection. This new information will be key for designing new ways to target risk reduction for recently HIV-infected men.

ELIGIBILITY:
Inclusion Criteria:

18 years of age or older Male Documented HIV infection that occurred within previous 12 months Willing to complete study procedures Mentally competent to give informed consent Willingness to refer partners to study Ability to complete practice questions for the web-based system

Exclusion Criteria:

Less than 18 years of age No report of sex with another man in the past 12 months

Unwilling to be tested for HIV including:

Unwilling to complete study follow-up questionnaires Not mentally competent to understand study procedures and give informed consent Unwilling to provide an email address or create one for the study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Study Population: STI/HIV testing and treatment clinic
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2009-02 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
To measure how HIV transmission risks change over time among recently HIV-infected individuals and their partners | 12 months
  This study will compare behavioral patterns of recently HIV infected individuals with those with chronic HIV infection and no HIV infection. It will allow for partnership level analyses by actively recruiting sexual partners.

CONTACTS AND LOCATIONS:
Overall Officials: Pamina M. Gorbach, DrPh, Principal Investigator — UCLA/EPI
Locations (1):
- Los Angeles Gay and Lesbian Center, Los Angeles, California, United States

REFERENCES:
- [Derived] Murray CH, Javanbakht M, Cho GD, Gorbach PM, Fulcher JA, Cooper ZD. Changes in Immune-Related Biomarkers and Endocannabinoids as a Function of Frequency of Cannabis Use in People Living With and Without HIV. Cannabis Cannabinoid Res. 2024 Jun;9(3):e897-e906. doi: 10.1089/can.2022.0287. Epub 2023 Apr 20. PMID 37093248
- See also: MetroMates Study Website — http://metromates.bol.ucla.edu/